CLINICAL TRIAL: NCT05716997
Title: A PRospective Observational Study on the Relationship BEtween Coronary Angiography Findings and Fractional Flow Reserve After Balloon Angioplasty: PROBE-FFR
Brief Title: Relationship Between Coronary Angiography Findings and Fractional Flow Reserve After Balloon Angioplasty
Acronym: PROBE-FFR
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: PROBE-FFR
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Fractional flow reserve; Balloon angioplasty; Coronary artery dissection; Coronary artery elastic recoil
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational study is to learn about in patients who need percutaneous coronary intervention for coronary artery disease. The main questions it aims to answer are:

* Fractional flow reserve according to coronary angiography findings after coronary artery balloon angioplasty
* Differences in fractional blood flow reserve before and after lesions between coronary balloon angioplasty using a scoring balloon and a regular balloon Participants will voluntarily consent to the study after being fully informed about the study and given ample opportunity to ask questions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically stable coronary artery disease
* Patients undergoing balloon angioplasty as an interventional procedure (FFR-guided PCI) using coronary artery fractional blood flow reserve for de novo lesions with a standard vessel diameter of 2.25 mm or more under percutaneous coronary angiography (hereafter referred to as coronary angiography)

(Note) If there are other lesions in the proximal area and the FFR of the distal lesion is collected, it is included in the selection target regardless of whether or not the proximal lesion was operated on.

Exclusion Criteria:

* Target lesion with stenosis of less than 50% or greater than 90% of the internal diameter
* Procedure for restenosis within the stent
* Pre-dilation performed on the target lesion before the coronary artery fractional blood flow reserve test
* Prior coronary artery bypass surgery
* Clinically unstable or ST-segment elevation myocardial infarction
* Myocardial infarction in the region supplied by the target vessel
* Target vessel is a blood vessel that supplies collateral circulation for occlusion of other blood vessels (not applicable when the need for collateral circulation has been resolved due to the opening of another vessel occlusion)
* Left ventricular ejection fraction (EF) less than 30%
* Most recently measured eGFR is less than 30 right before the procedure
* Accompanying primary valve disease requiring treatment
* Accompanying primary heart disease such as dilated cardiomyopathy, hypertrophic cardiomyopathy, or restrictive cardiomyopathy
* Congenital heart disease

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met the inclusion criteria and underwent interventions, as determined by clinical necessity, using fractional blood flow reserve (FFR) after percutaneous coronary angiography (PCA) will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Differences in fractional flow reserve (FFR) according to angiographic findings after coronary artery balloon angioplasty | 15 minutes
  Coronary angiographic findings and fractional flow within 15 minutes after coronary balloon angioplasty are collected and analyzed.

SECONDARY OUTCOMES:
Comparison of differences in fractional flow reserve (FFR) before and after lesions between coronary balloon angioplasty using a scoring balloon and a regular balloon | 1 year
  Determine whether a scoring balloon or a general balloon was used during balloon angioplasty, and analyze whether there is a difference in FFR depending on the balloon used.
1-year outcome | 1 year
  Relationship between major cardiac events within 1 year according to changes in pre- and post-lesional fractional flow reserve (FFR), steady-state pressure ratio, and quantitative flow analysis (QFR) values before and after coronary artery balloon angioplasty
Relationship between fractional blood flow reserve and intravascular ultrasound lesion-specific minimum lumen area | 1 year
  Relationship between fractional blood flow reserve and intravascular ultrasound lesion-specific minimum lumen area (mm2)
Relationship between fractional blood flow reserve and intravascular ultrasound lesion-specific plaque burden | 1 year
  Relationship between fractional blood flow reserve and intravascular ultrasound lesion-specific plaque burden (plaque burden = plaque cross-sectional area (CSA, mm2)+ media CSA / external elastic membrane CSA)
Relationship between fractional blood flow reserve and intravascular ultrasound lesion-specific positive remodeling | 1 year
  Relationship between fractional blood flow reserve and intravascular ultrasound lesion-specific positive remodeling (remodeling ratio > 1.05).
  remodeling ratio (RR) = external elastic membrane (EEM) area lesion/EEM area proximal reference
Relationship between fractional blood flow reserve and intravascular ultrasound lesion-specific attenuated plaque | 1 year
  Relationship between fractional blood flow reserve and intravascular ultrasound lesion-specific attenuated plaque Attenuated Plaque: Plaque seen in intravascular ultrasound with acoustic shadowing behind large, echolucent acute culprit lesion sites, in the absence of bright calcium.

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, Study Chair — Seoul National University Hospital; Bon-Kwon Koo, MD, Study Director — Seoul National University Hospital; Bon-Kwon Koo, MD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Ewha Womans University Mokdong Hospital, Seoul
  - Seou National University Hospital, Seoul